CLINICAL TRIAL: NCT04778709
Title: A Randomized, Split Mouth Study of the Effects of Bone Graft Particle Size on Bone Vitality and Bone Volume Outcomes in Subjects Undergoing Sinus Augmentation for the Placement of Dental Implants
Brief Title: Bone Graft Particle Size on Bone Vitality and Volume
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI who is no longer at the institution, the sponsor of this research study, Zimmer Biomet, along with the current PI have decided to close enrollment to the study and to early terminate the study.
Sponsor: NYU College of Dentistry (Other)
Responsible Party: Principal Investigator, Katerina Georgantza, DDS, Clinical Assistant Professor, NYU College of Dentistry
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19-00996
Record Dates: First submitted 2021-01-30; First posted 2021-03-03 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bilateral Sinus Pneumatization; Posterior Maxillary Ridge Atrophy Due to Extraction
Keywords: Sinus floor augmentation; Bone graft; Allograft; Dental implants; Maxillary sinus

STUDY DESIGN:
Intervention Model Description: Each subject will receive bilateral sinus augmentation. Right and left sinuses will be randomly assigned to Bone Graft A and Bone Graft B.
Who Masked: Participant, Outcomes Assessor
Masking Description: CBCT review, core biopsy evaluation and histomorphometry will be performed by a masked investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bone Graft A (Experimental): Bone Graft A: Mixture of 25% small-particle cortical, 25% large particle cortical, 25% small particle cancellous, 25% large particle cancellous allograft
  Interventions: Device: Puros allograft
- Bone Graft B (Active Comparator): Bone Graft B: 100% large particle cancellous allograft
  Interventions: Device: Puros allograft

INTERVENTIONS:
Device: Puros allograft — Bilateral sinus augmentation procedure using the lateral window technique. Graft material combination A or B will be randomly assigned to right and left sinus.
  Each subject will receive the following bone allograft material:
  Four to six grams of commercially available human donor bone allograft (Puros Allograft Bone Particles, Zimmer Biomet, Palm Beach Gardens, FL USA) consisting of Graft A cortical and cancellous bone chips of both 250-1000 microns and 1000-2000 microns size, or Graft B for contralateral sinus: cancellous 1000-2000 microns size alone.

SUMMARY:
To determine the effects of small and large bone graft particles vs large particles alone on percent vital bone, percent residual graft material, measured histologically from bone biopsies of the grafted site taken at the time of dental implant placement from subjects undergoing sinus augmentation for the placement of dental implants. Dental radiographs taken post operatively will be used to estimate bone graft volume differences between conditions.

DETAILED DESCRIPTION:
The proposed study is a Randomized, single-masked, split-mouth, single center study.

About 20 subjects will be screened in order to randomize 10 study subjects. 10 patients who needing bilateral sinus augmentation procedure using the lateral window technique will be randomized using computer generated randomized technique.

At the day of the surgical procedure each tooth sites will be randomized 1:1 into one of the following bone grafts to either the right or left side of the mouth.:

* Bone graft A: A mixture of 25% small-particle cortical allograft, 25% large-particle cortical allograft, 25% small-particle cancellous allograft, and 25% large-particle cancellous allograft is used for one sinus (N=10)
* Bone graft B: 100% large particle cancellous allograft for the contralateral sinus (N=10) Immediately after the sinus augmentation surgery a CBCT will be acquired and will be compared to a second CBCT prior to implant placement in order to compare the volumetric changes in the sinus.

At the visit of implant placement, a bone core will be collected from both sinuses for histomorphometric evaluation to evaluate the residual graft particles, the new vital bone formation and the amount of soft tissue components.

ELIGIBILITY:
Inclusion Criteria:

* Good physical health
* Capable of maintaining good oral hygiene
* Missing posterior maxillary teeth on both sides and less than 5 mm of residual jaw bone requiring maxillary sinus augmentation prior to dental implant placement
* Capable and willing to give informed consent

Exclusion Criteria:

* The presence of underlying medical conditions that may pose an undue risk for sinus surgery
* Patients with untreated oral infections
* Pregnant and lactating females
* Individuals who have the habit of smoking and/or tobacco chewing
* Patients not willing to participate in the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Implant Dentistry, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: tooth sites
Groups:
- Bone Graft A: Bone Graft A: Mixture of 25% small-particle cortical, 25% large particle cortical, 25% small particle cancellous, 25% large particle cancellous allograft
  Puros allograft: Bilateral sinus augmentation procedure using the lateral window technique. Graft material combination A or B will be randomly assigned to right and left sinus.
  Each subject will receive the following bone allograft material:
  Four to six grams of commercially available human donor bone allograft (Puros Allograft Bone Particles, Zimmer Biomet, Palm Beach Gardens, FL USA) consisting of Graft A cortical and cancellous bone chips of both 250-1000 microns and 1000-2000 microns size, or Graft B for contralateral sinus: cancellous 1000-2000 microns size alone.
- Bone Graft B: Bone Graft B: 100% large particle cancellous allograft
  Puros allograft: Bilateral sinus augmentation procedure using the lateral window technique. Graft material combination A or B will be randomly assigned to right and left sinus.
  Each subject will receive the following bone allograft material:
  Four to six grams of commercially available human donor bone allograft (Puros Allograft Bone Particles, Zimmer Biomet, Palm Beach Gardens, FL USA) consisting of Graft A cortical and cancellous bone chips of both 250-1000 microns and 1000-2000 microns size, or Graft B for contralateral sinus: cancellous 1000-2000 microns size alone.
Period: Overall Study
Arm/Group | Bone Graft A | Bone Graft B
Started | 2; 4 tooth sites | 2; 4 tooth sites
Completed | 0; 0 tooth sites | 0; 0 tooth sites
Not Completed | 2; 4 tooth sites | 2; 4 tooth sites

BASELINE CHARACTERISTICS:
Units Other Than Participants: Tooth Sites
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Graft A | Bone Graft B | Total
Number analyzed (Participants) | 2 | 2 | 4
Number analyzed (Tooth Sites) | 4 | 4 | 8
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 0 | 0 | 0
  26-35 years | 0 | 0 | 0
  36-45 years | 0 | 0 | 0
  46-55 years | 0 | 0 | 0
  56-65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 1
  Non-Hispanic White | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Quality of Bone
Description: Assessment of the quality of bone that is generated in the grafted sinuses by measuring the: percent vital bone formation, percent of inflammatory tissue if any
Time Frame: After surgery, 8 months, 1 year
Population: Data were not collected. The original PI who is no longer at the institution, the sponsor of this research study, Zimmer Biomet, along with the current PI has decided to close enrollment to the study and to early terminate the study.
Arm/Group | Bone Graft A | Bone Graft B
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Quality of Bone
Description: Assessment of the quality of bone that is generated in the grafted sinuses by measuring the: percent of residual bone graft material
Time Frame: After surgery, 8 months, 1 year
Population: as for outcome 1
Arm/Group | Bone Graft A | Bone Graft B
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Quality of Bone
Description: Assessment of the quality of bone that is generated in the grafted sinuses by measuring the: percent of inflammatory tissue if any
Time Frame: After surgery, 8 months, 1 year
Population: as for outcome 1
Arm/Group | Bone Graft A | Bone Graft B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Bone Volume Stability
Description: Assessment of bone volume stability through CBCT analysis comparing it from the time of placement, 8 months post-grafting and 1 year post-implantation
Time Frame: After surgery, 8 months, 1 year
Population: as for outcome 1
Arm/Group | Bone Graft A | Bone Graft B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 months
Description: Data on all serious and non-serious Adverse Events experienced by participants were collected, irrespective of the event's relation to the tooth site.
Arm/Group | Bone Graft A | Bone Graft B
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT04778709/Prot_SAP_000.pdf